CLINICAL TRIAL: NCT01956721
Title: Evaluation of Calcium Homeostasis and Mitochondrial Function in Skeletal Muscle in Subjects With Heart Failure
Brief Title: Impact of Heart Failure on Calcium Homeostasis and Mitochondrial Function in Human Skeletal Muscle
Acronym: CALCICARD2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty of inclusion
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Ministry of Health, France (Other Government); National Cancer Institute, France (Other Government); Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9051
Record Dates: First submitted 2013-06-12; First posted 2013-10-08 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure
Keywords: Heart Failure , Skeletal muscle,Calcium,Ryanodine Receptor, Mitochondria, Exercise training, Muscle biopsy, Healthy volunteers
MeSH Terms: conditions — Heart Failure | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Patients with heart failure (FEVG ≥ 50%) (Experimental): Patients with heart failure (FEVG ≥ 50%)
  Interventions: Procedure: Exercise training,; Procedure: Muscle biopsy
- Patients with heart failure (FEVG ≤ 35%), (Experimental): Patients with heart failure (FEVG ≤ 35%),
  Interventions: Procedure: Exercise training,; Procedure: Muscle biopsy
- Healthy Volunteers (Other): Healthy Volunteers with no heart failure
  Interventions: Procedure: Exercise training,; Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Exercise training,
Procedure: Muscle biopsy

SUMMARY:
The aim of this project is to investigate the impact of heart failure (HF) on calcium homeostasis, mitochondrial function and oxydative stress in human skeletal muscle. The role playing by circulating factors such as cytokines and catecholamines will also be evaluated. 24 HF patients wiil be enrolled in the study: 12 male volunteers with a fraction of ejection ≥ 50% and 12 male volunteers with a fraction of ejection ≤ 35%. They will be compared to 12 sedentary healthy male volunteers, matched on age and physical activity.

DETAILED DESCRIPTION:
Heart Failure ( HF) is associated with a skeletal muscle dysfunction, characterized by an increased fatigue that does not correlate with impaired myocardial function and physical inactivity that is commonly associated with HF. We identified in skeletal muscle of HF rats, a dysfunction of type 1 ryanodine receptors (RyR1) similar to that observed on the cardiac channel ( RyR2), due to an hyperphosphorylation of the RyR and a dissociation of the regulatory protein FKBP12. This dysfunction, in addition to mitochondrial impairment, contributes in this animal model to the reduced exercise capacity observed during HF. Our goal is to analyse the impact of HF on calcium homeostasis, mitochondrial function and oxydative stress in human skeletal muscle. This project, performed on muscle biopsies, will also allow us to correlate calcium homeostasis and mitochondrial function to circulating factors ( cytokines, catecholamines) susceptible to trigger this muscle dysfunction.This project addresses two straightforward questions about physiopathological mechanisms involved in skeletal muscle dysfunction during HF. To this aim we have built locally a network of laboratories and clinical services, used to work together, composed of two services of the University Hospital of Montpellier ( Dept. of Cardiology and Dept of Clinical Physiology), an inserm unit (U1046, team 2) all interfaced by an another Inserm facility: the Clinical Investigation center (CIC) of Montpellier. In this project we will focus on the dilated post-ischemic cardiomyopathy and compare two groups of patients under similar treatments studied at different stages of HF. The first patients with a fraction of ejection ≥ 50% will be compares with patients) with an ejection fraction ≤ 35% (12 males, 35-65 years old per HF). 12 voluntary healthy sedentary individuals carefully selected for similar level of activity as for patients will be matched to the HF groups. All individuals will undergo cardiovascular explorations (ECG and echocardiography, blood test) at the inclusion. They will perform an exercise testing to evaluate their exercise capacity. A muscle biopsy will be performed between 4 and 8 days after the exercise testing to assess the mitochondrial function and the Ca2+ homeostasis. This project will allow us to characterize the behavior of RyR in relation with mitochondrial function in human skeletal muscle during HF . The analysis of circulating factors will allow us to establish a relation of cause and effect between myocardial dysfunction and muscle dysfunction. This project could thus open important perspectives in therapeutic. Compounds analogues to JTV-519, acting in stabilizing RyR channels, could be prescribed as a potent medication for HF. This project could thus be determinant in the comprehension of the regulation of Ca2+ and energetic metabolism in human skeletal muscle which could be an appropriate model to evaluate the effects of new pharmacological agents.

ELIGIBILITY:
Inclusion Criteria:

* - BMI < 30

Exclusion Criteria:

* Contra-indication to exercise testing performance and muscle biopsy

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-09-18 (Actual); Primary Completion 2016-06-21 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
calcium homeostasis | 8 days
  Cell analysis
mitochondrial function | 8 days
  Cell analysis

SECONDARY OUTCOMES:
skeletal muscular function in two stages of heart failure | 8 days
  Cell analysis

CONTACTS AND LOCATIONS:
Locations (1):
- physiologie clinique, hopital Arnaud de Villeneuve, 371 avenue du Doyen G;Giraud, Montpellier, France